CLINICAL TRIAL: NCT01982383
Title: A Prospective Study of the Use of Micropulse 577nm Laser Treatment in Central Serous Chorioretinopathy
Brief Title: Study on the Use of Micropulse Laser to Treat Central Serous Chorioretinopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 021236
Record Dates: First submitted 2013-11-06; First posted 2013-11-13 (Estimated); Results first posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Central Serous Chorioretinopathy
Keywords: CSC; Edema; Retinopathy
MeSH Terms: conditions — Central Serous Chorioretinopathy; Edema; Retinal Diseases | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micropulse Laser Treatment (Experimental): Patient's randomized to ML treatment would be treated with the following settings: 200 micron spot size, 0.2 second duration, 15% duty cycle, and 300 milliWatt power. Their eyes would be dilated prior to treatment with standard mydriatic medications, including Tropicamide and Phenylephrine
  Interventions: Device: Micropulse Laser Treatment
- No Treatment (Placebo Comparator): Patients randomized to this treatment arm, will not receive treatment for CSC. They will continue to be observed at month 1 and month 3. If any worsening of pathology is found during the follow up visits, the patient will be removed from the study and given appropriate standard of care by the attending
  Interventions: Other: No treatment

INTERVENTIONS:
Device: Micropulse Laser Treatment
  Other Names: Micropulse 577nm; Laser
  Arms: Micropulse Laser Treatment
Other: No treatment
  Arms: No Treatment

SUMMARY:
The investigators hypothesis is that using the micropulse laser in patient with Central Serous Chorioretinopathy (CSC) will prompt resolution of CSC and will be effective in significantly minimizing visual recovery time from this disease as well as potentially preventing recurrences.

DETAILED DESCRIPTION:
The investigators hypothesize that application of 577nm micropulse laser in patients with CSC will prompt resolution of CSC as measured by ocular coherence tomography and best corrected visual acuity. This will be a pilot study to establish sound methods and provide some insights to the safety and efficacy of CSC treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with new diagnosis of CSC and no other comorbidities or prior retinal treatment
* Patients ranging from 30 to 60 years of age

Exclusion Criteria:

* Patients with no case of CSC
* Patients with other macular comorbidities including but not limited to diabetic retinopathy, macular degeneration
* Patients with prior retinal treatment

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2012-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeevan Mathura, MD, Principal Investigator — George Washington University
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Ricci F, Missiroli F, Cerulli L. Indocyanine green dye-enhanced micropulsed diode laser: a novel approach to subthreshold RPE treatment in a case of central serous chorioretinopathy. Eur J Ophthalmol. 2004 Jan-Feb;14(1):74-82. doi: 10.1177/112067210401400115. PMID 15005592
- [Background] Lanzetta P, Furlan F, Morgante L, Veritti D, Bandello F. Nonvisible subthreshold micropulse diode laser (810 nm) treatment of central serous chorioretinopathy. A pilot study. Eur J Ophthalmol. 2008 Nov-Dec;18(6):934-40. doi: 10.1177/112067210801800613. PMID 18988165
- [Background] Chen SN, Hwang JF, Tseng LF, Lin CJ. Subthreshold diode micropulse photocoagulation for the treatment of chronic central serous chorioretinopathy with juxtafoveal leakage. Ophthalmology. 2008 Dec;115(12):2229-34. doi: 10.1016/j.ophtha.2008.08.026. PMID 19041477
- [Derived] Lange CA, Qureshi R, Pauleikhoff L. Interventions for central serous chorioretinopathy: a network meta-analysis. Cochrane Database Syst Rev. 2025 Jun 16;6(6):CD011841. doi: 10.1002/14651858.CD011841.pub3. PMID 40522203

RESULTS

PARTICIPANT FLOW:
Groups:
- Micropulse Laser Treatment: Patient's randomized to ML treatment would be treated with the following settings: 200 micron spot size, 0.2 second duration, 15% duty cycle, and 300 milliWatt power. Their eyes would be dilated prior to treatment with standard mydriatic medications, including Tropicamide and Phenylephrine
  Micropulse Laser Treatment
- No Treatment: Patients randomized to this treatment arm, will not receive treatment for CSC. They will continue to be observed at month 1 and month 3. If any worsening of pathology is found during the follow up visits, the patient will be removed from the study and given appropriate standard of care by the attending
  No treatment
Period: Overall Study
Arm/Group | Micropulse Laser Treatment | No Treatment
Started | 2 | 0
Completed | 2 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Micropulse Laser Treatment | No Treatment | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Fluid Build-up
Description: Central Serous Choroidopathy is a disease that causes fluid to build up under the retina,the back part of the inner eye that sends sight information to the brain. The objective here is to apply 577nm of micropulse laser to see if CSC resolution occurs and measuring it through ocular coherence tomography (retinal imaging), vision score, and visual field testing for retinal sensitivity.
Time Frame: within 1 week to 3 months after the laser procedure is completed
Population: No data analyzed. Study terminated due to lack of enrollment
Arm/Group | Micropulse Laser Treatment | No Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Micropulse Laser Treatment | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes